CLINICAL TRIAL: NCT00609505
Title: Telemedicine vs. Face-to-Face Cancer Genetic Counseling in Rural Oncology Clinics
Brief Title: Telemedicine vs. Face-to-Face Cancer Genetic Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00001547; DISP0707781
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Hereditary Breast and Ovarian Cancer Syndrome; Lynch Syndrome
Keywords: Hereditary Breast and Ovarian Cancer syndrome; genetic counseling; breast cancer; ovarian cancer; telemedicine; Cancer genetic counseling
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome; Colorectal Neoplasms, Hereditary Nonpolyposis; Breast Neoplasms; Ovarian Neoplasms | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TM (Other): Telemedicine genetic counseling group
  Interventions: Other: Telemedicine
- FTF (Other): Face-to-face genetic counseling group
  Interventions: Other: Face-to-Face

INTERVENTIONS:
Other: Telemedicine — Telemedicine genetic counseling
  Arms: TM
Other: Face-to-Face — Face-to-face genetic counseling
  Arms: FTF

SUMMARY:
Cancer genetic counseling (CGC) has been found to have "substantial" benefits for individuals with breast cancer and their family members; it has been deemed by multiple organizations as "standard of care" for women with breast cancer and their relatives. Unfortunately, there is a disparity in access to CGC, especially among women who live in rural and underserved areas. In North Carolina, only two cancer genetic counselors practice in rural clinics - each only for a few days per month. Therefore, in an effort to make CGC more widely available in a timely manner, we propose to test provision of counseling through telemedicine (TM), in which a patient and health care provider communicate with each other using videoconferencing. In 4 rural oncology clinics, we will implement low-cost TM and compare satisfaction and cost-effectiveness between groups of women designated to have their CGC session by TM or FTF. We'll use a validated measure to assess satisfaction by a phone survey one week after the CGC appointment; cost-effectiveness will be measured at project's end by calculating length of wait time for appointment and costs of equipment, labor, and mileage. Study hypothesis: TM is as satisfactory as FTF counseling and is a more cost-effective way to provide this beneficial service.

ELIGIBILITY:
Inclusion Criteria:

* Individuals referred for cancer genetic counseling (e.g., by medical oncologist, primary care physician or self) in one of 4 oncology clinics: Gibson Cancer Center in Lumberton, NC; Scotland Cancer Treatment Center in Laurinburg, NC; Johnston Cancer Center in Smithfield, NC; and Maria Parham Cancer Center in Henderson, NC.
* Willing to be randomized to receive counseling via telemedicine or face-to-face.

Exclusion Criteria:

* Referred for cancer genetic counseling from any clinic other than the 4 listed above.
* Unwilling to be randomized to receive counseling via telemedicine or face-to-face.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-08; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | One week post-intervention (genetic counseling session)

SECONDARY OUTCOMES:
Cost-effectiveness | Enrollment completion

CONTACTS AND LOCATIONS:
Overall Officials: Martha B Adams, M.D., M.A., Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Maria Parham Medical Center, Henderson, North Carolina
  - Scotland Cancer Treatment Center, Laurinburg, North Carolina
  - Gibson Cancer Center, Lumberton, North Carolina
  - Johnston Cancer Center, Smithfield, North Carolina

REFERENCES:
- [Derived] Buchanan AH, Datta SK, Skinner CS, Hollowell GP, Beresford HF, Freeland T, Rogers B, Boling J, Marcom PK, Adams MB. Randomized Trial of Telegenetics vs. In-Person Cancer Genetic Counseling: Cost, Patient Satisfaction and Attendance. J Genet Couns. 2015 Dec;24(6):961-70. doi: 10.1007/s10897-015-9836-6. Epub 2015 Apr 3. PMID 25833335
- See also: Duke Hereditary Cancer Clinic website — http://www.dukehealth.org/Services/HereditaryCancer/index
- See also: Duke Oncology Network website — http://www.cancer.duke.edu/don/